CLINICAL TRIAL: NCT06736301
Title: An Exploratory Clinical Study of Double Pig Tail Stent-assisted Fixation of Fully Covered Metal Stents for the Treatment of Benign Duodenal Strictures
Brief Title: Double Pig Tail Stent-assisted Fixation of Fully Covered Metal Stents for the Treatment of Benign Duodenal Strictures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shupei Li (Other)
Responsible Party: Sponsor-Investigator, Shupei Li, student, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLL-24-40
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Benign Duodenal Stricture
Keywords: duodenal stricture; fully covered stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stent (Experimental): a double pig-tail stent for cross fixation of a fully covered stent
  Interventions: Device: a fully covered stent

INTERVENTIONS:
Device: a fully covered stent — a double pig-tail stent for cross fixation of a fully covered stent

SUMMARY:
Double Pig Tail Stent-assisted Fixation of Fully-Covered Metal Stents for the Treatment of Benign Duodenal Strictures

DETAILED DESCRIPTION:
This study uses a double pig-tail stent for cross fixation of a fully-covered stent in the duodenum to reduce the incidence of displacement and ensure the stent can effectively expand the narrowed area, thereby alleviating patient symptoms.

The aim of this study is to explore the safety and efficacy of a double pig-tail stent-assisted fixation of a fully-covered stent for the treatment of benign duodenal strictures, further clarifying its long-term efficacy and providing strong support for the placement of fully-covered stents in treating benign duodenal strictures.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily signed the informed consent form for this trial;
2. Patients diagnosed with benign duodenal stricture;
3. Symptoms of upper gastrointestinal obstruction, such as nausea, vomiting, abdominal pain, or changes in bowel habits, occurring before admission or during hospitalization;
4. Patients with refractory strictures who have failed multiple balloon dilations;
5. Age < 75 years.

Exclusion Criteria:

1. Gastrointestinal perforation;
2. Distal small bowel obstruction or multiple segments of small bowel obstruction;
3. Coagulation disorders;
4. Strictures or obstructions caused by malignant tumors;
5. Severe comorbidities involving the heart, brain, lungs, kidneys, etc.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate at 30 days post-operation | at 30 days post-operation
  Clinical remission: Symptoms of duodenal obstruction are relieved, and the postoperative GOOSS score improves by at least one grade compared to preoperative values.

CONTACTS AND LOCATIONS:
Locations (1):
- Fully Covered Metal Stents, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No